CLINICAL TRIAL: NCT05904587
Title: Clinical Evaluation of the Effectiveness of Different Methods in Reducing Pain During Debonding of Orthodontic Fixed Appliance: a Randomized Clinical Trial
Brief Title: Methods That Reduce Pain During Debonding Fixed Orthodontic Appliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Alhasan Ibraheem Ali, B.D.S., University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 780423
Record Dates: First submitted 2023-06-04; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pain
Keywords: pain and debonding
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- open mouth debonding (No Intervention): debonding of the bracket is done while the mouth of the patient is open and without any support to the teeth during the debonding procedure
- biting on soft elastomeric wafer (Experimental): debonding of the bracket is done while the patient is biting on the preshaped soft elastomeric wafer (cut into a horseshoe shape) during the debonding procedure
  Interventions: Other: ortho technology, sports advantage, thermal forming soft EVA 3mm
- biting on cotton roll (Experimental): debonding of the bracket is done while the patient is biting on a cotton roll during the debonding procedure
  Interventions: Other: cotton roll
- biting on the mouthpiece of vibrational device (Experimental): debonding of the bracket is done while the patient is biting on the mouthpiece of the vibrational device (SureSmile® VPro™) delivering vibrations to the dentition during the debonding procedure
  Interventions: Device: SureSmile® VPro™

INTERVENTIONS:
Device: SureSmile® VPro™ — the pain is recorded when the patient is biting on the mouthpiece of the device during the debonding procedure
  Arms: biting on the mouthpiece of vibrational device
Other: ortho technology, sports advantage, thermal forming soft EVA 3mm — the pain is recorded when the patient is biting on the EVA sheet during the debonding procedure
  Arms: biting on soft elastomeric wafer
Other: cotton roll — the pain is recorded when the patient is biting on the cotton roll during the debonding procedure
  Arms: biting on cotton roll

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of four different methods (including the control group) in reducing pain during debonding of fixed orthodontic appliances in participants requiring the removal of their fixed orthodontic appliance.

The main question it aims to answer is which method (biting on a cotton roll, biting on a soft thermoplastic elastomeric sheet, and the use of low-level vibration in reducing pain during the debonding procedure) is most effective in reducing the patients' pain during debonding of conventional orthodontic fixed appliances.

Participants will be asked to give their pain score on a scale of 0 to 100 VAS (visual analogue scale) for every region of the dentition.

the researcher then will compare different scores of different methods to find the most effective method in reducing pain.

DETAILED DESCRIPTION:
After signing the consent form, the patient will be tested using General Anxiety Disorder 7 (GAD-7) to reduce the effect of general anxiety on pain scores. GAD consists of 7 statements designed to measure anxiety. This will aid in identifying individuals who have severe anxiety disorder and exclude them from the study to ensure more accurate results.

Four debonding methods will be used in this study; Routine mechanical debonding with debonding plier with an open mouth, which will be used as control, and three other interventions to manage pain including biting on a cotton roll, biting on an elastomeric wafer, and using vibration. All of the procedures will be done with the archwire in situ and with minimal torsional force on the bracket.

For the control group, the debonding will be done with an open-mouth technique without any support applied to the teeth. The cotton roll method will be done by asking the patient to bite on the cotton roll firmly but not excessively during the debonding procedure.

As for the elastomeric wafer group the patient will bite on the wafer firmly during the debonding procedure, in a similar fashion the patient will bite on the mouthpiece of the VPro vibration device.

Pain will be estimated by using 100mm VAS and recording the results for each sextant, accompanied by the GAD-7 results and the patient's age and gender.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between 15-30 years of age who could understand, assess, and answer the questionnaires.
2. No history of taking medicine periodically or in the last 24 hours (e.g., painkillers, corticosteroids, and anti-flu drugs).
3. No debonded brackets prior to debonding procedure.
4. No missing teeth except extracted premolar.
5. Undergoing upper and lower fixed orthodontic treatment with 0.022-inch metal brackets.
6. Finishing arch wires present for at least two months.
7. No craniofacial deformities that would affect the dentoalveolar bone quality (e.g., cleft lip and palate) .

Exclusion Criteria:

1. History of taking medicine periodically or in the last 24 h (e.g., analgesic, anti-inflammatory and anxiolytic).
2. GAD-7 score of ˃8.
3. Debonded brackets at the time of debonding.
4. Missing teeth except for extracted premolars.
5. Active periodontal problems (recession and mobility greater than Grade I),
6. Heavily restored or root canal treated tooth.
7. Craniofacial deformities that would affect dentoalveolar bone quality (e.g., cleft lip and palate).
8. Surgical treatment (including impacted tooth removal) and presence of mini-screws.
9. excessive gingival overgrowth.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-03-19 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
pain during debonding of conventional fixed orthodontic appliance | Intraprocedural
  pain will be estimated using 0-100 VAS (visual analogue scale) of each segment of the dentition during the debonding procedure

SECONDARY OUTCOMES:
the dentition segment with the highest pain scores | Intraprocedural
  will be measured statistically

CONTACTS AND LOCATIONS:
Overall Officials: Ammar S Kadhum, Asst. Prof., Study Director — University of Baghdad
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Bab Al-Muadham, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with an academic interest in pain and debonding of conventional fixed orthodontic appliances. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)

REFERENCES:
- [Background] Almuzian M, Rizk MZ, Ulhaq A, Alharbi F, Alomari S, Mohammed H. Effectiveness of different debonding techniques and adjunctive methods on pain and discomfort perception during debonding fixed orthodontic appliances: a systematic review. Eur J Orthod. 2019 Sep 21;41(5):486-494. doi: 10.1093/ejo/cjz013. PMID 30934051
- [Background] Bavbek NC, Tuncer BB, Tortop T, Celik B. Efficacy of different methods to reduce pain during debonding of orthodontic brackets. Angle Orthod. 2016 Nov;86(6):917-924. doi: 10.2319/020116-88R.1. Epub 2016 May 12. PMID 27172508
- [Background] Celebi, F. (2021) Evaluation of the effects of cotton roll-biting on debonding pain: a split-mouth study. South European Journal of Orthodontics And Dentofacial Research, 8, 1-7.
- [Background] Gupta SP, Rauniyar S, Prasad P, Pradhan PMS. A randomized controlled trial to evaluate the effectiveness of different methods on pain management during orthodontic debonding. Prog Orthod. 2022 Mar 1;23(1):7. doi: 10.1186/s40510-022-00401-y. PMID 35229220
- [Background] Jaypapal, J., Maheshwari, U. and Vijayalakshmi, V. (2020) Comparison of pain perception during debonding between conventional and vibratory therapy. Annals of the Romanian Society for Cell Biology, 24, 701-715.
- [Background] Kilinc DD, Sayar G. Evaluation of pain perception during orthodontic debonding of metallic brackets with four different techniques. J Appl Oral Sci. 2019 Jan 7;27:e20180003. doi: 10.1590/1678-7757-2018-0003. PMID 30624460
- [Background] Pithon MM, Santos Fonseca Figueiredo D, Oliveira DD, Coqueiro Rda S. What is the best method for debonding metallic brackets from the patient's perspective? Prog Orthod. 2015;16:17. doi: 10.1186/s40510-015-0088-7. Epub 2015 Jun 17. PMID 26081783
- [Background] Williams OL, Bishara SE. Patient discomfort levels at the time of debonding: a pilot study. Am J Orthod Dentofacial Orthop. 1992 Apr;101(4):313-7. doi: 10.1016/S0889-5406(05)80324-5. PMID 1558060
- [Derived] Musawi AI, Kadhum AS. Effectiveness of high-frequency vibration, cotton rolls and elastomeric wafers in alleviating debonding pain of orthodontic metal brackets: a randomized clinical trial. Sci Rep. 2024 Oct 24;14(1):25160. doi: 10.1038/s41598-024-75725-2. PMID 39448724